CLINICAL TRIAL: NCT04853212
Title: The Role of Dysbiosis of Intestinal Microbiota in the Development of Spondyloarthritis
Brief Title: The Role of Intestinal Microbiota Dysbiosis in the Development of Spondyloarthritis
Acronym: RUMINOSPA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP210332; 2020-A03244-35 (Registry Identifier: IDRCB)
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Spondyloarthritis; Ruminococcus Gnavus
Keywords: Spondyloarthritis; Ruminococcus gnavus; Microbiota; Dysbiosis
MeSH Terms: conditions — Spondylarthritis; Dysbiosis | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPA patient (Active Comparator): Patients with SPA
  Interventions: Procedure: Biopsy
- Subject without SPA (Sham Comparator): Health subjects without SPA, planned to undergo a digestive endoscopy.
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — Biopsy during recto-coloscopy

SUMMARY:
The primary objective of this case-control study aims to explore the role of bacterium Ruminococcus gnavus (R. gnavus) with intestinal biopsy and faecal sampling in the initiation and the development of spondyloarthritis (SPA) in comparison with health control subjets (patients without chronic disease but have indication to digestive endoscopy).

DETAILED DESCRIPTION:
As secondary objectives, the study aims:

* to research the abundance of bacterial strain of R. gnavus in mucosal sampling by biopsy;
* to study the interaction between R. gnavus bacterium and mucus from histological sampling;
* to correlate the expression of genes of intestinal mucus with the variations of identified microbiota of mucus biopsy;
* to study the interaction between bacteria and intestinal epithelial cells during culture;
* to demonstrate perturbations of the immune responses by dysbiosis.

ELIGIBILITY:
Inclusion Criteria:

Patients with SPA:

* Patients ⩾ 18 years;
* Diagnosed as spondyloarthritis (SpA) according ASAS classification;
* Affiliated to a social security scheme;
* Have signed the written informed consent form.

Control subjects:

* Subjects ⩾ 18 years;
* Subjects free of SPA and planned for a digestive endoscopy for another indication such as to explore the risk of colorectal cancer in family member;
* Affiliated to a social security scheme;
* Have signed the written informed consent form.

Exclusion Criteria:

* Subjects unable to understand the proposed study and/or sign a informed consent form;
* Pregnant women or breast feeding women;
* Subjects under guardianship or curatorship;
* Have taken antibiotic 1 month prior to inclusion;
* Presenting acute or chronic severe pathology may likely to interfere with the interpret of outcome;
* Refusal of subjects to participate to the study;
* Foreign patients under french AME scheme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06-14 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Isolation and characterization of R. gnavus | At the end of study, up to 2 years
  Isolation and characterization of R. gnavus bacterium from intestinal biopsy.
Bacteria analysis | At the end of study, up to 2 years
  Analysis of repartition of R. gnavus bacterium in each group and the comparison between 2 groups.

SECONDARY OUTCOMES:
Bacterial strain's abundance | At the end of study, up to 2 years
  Compare the abundance by RT-q-PCR of bacterial strain (R. gnavus) between mucus biopsy sampling and faecal sampling, collected from PCR patients or control subjects respectively.
Mucin-degradation of Ruminococcus gnavus | At the end of study, up to 2 years
  Study the ability of the strain to grow on mucins of intestinal biopsy, colored after fixation to carnoy.
RNA sequencing analysis of biopsy | At the end of study, up to 2 years
  RNA sequencing analysis of rectal biopsy between SPA patients and control subjects.
Interaction between bacteria and intestinal epithelial cells | At the end of study, up to 2 years
  In order to study the interaction between bacteria and intestinal epithelial cells in culture (organoids).
  Study the induction of several target genes as peptides anti-microbians, mucin or chemokines by RT-q-PCR.
Dysbiosis-induced immune perturbations | At the end of study, up to 2 years
  To compare between 2 groups their reactivities of T cells from intestinal biopsy which contact with cells of exposed antigens in vitro, to R. gnavus stains or to other stains biopsied from control subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Maxime BREBAN, MD, PhD, Principal Investigator — Service de Rhumatologie, Hôpital Ambroise Paré, APHP
Locations (1):
- Service de Rhumatologie, Hôpital Ambroise Paré, APHP, Boulogne-Billancourt, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Breban M, Tap J, Leboime A, Said-Nahal R, Langella P, Chiocchia G, Furet JP, Sokol H. Faecal microbiota study reveals specific dysbiosis in spondyloarthritis. Ann Rheum Dis. 2017 Sep;76(9):1614-1622. doi: 10.1136/annrheumdis-2016-211064. Epub 2017 Jun 12. PMID 28606969
- [Background] Crost EH, Tailford LE, Monestier M, Swarbreck D, Henrissat B, Crossman LC, Juge N. The mucin-degradation strategy of Ruminococcus gnavus: The importance of intramolecular trans-sialidases. Gut Microbes. 2016 Jul 3;7(4):302-312. doi: 10.1080/19490976.2016.1186334. Epub 2016 May 25. PMID 27223845